CLINICAL TRIAL: NCT00305006
Title: Bimanual Training (HABIT) in Children With Hemiplegic Cerebral Palsy
Brief Title: Constraint-induced Movement Therapy (CIMT) and Bimanual Training (HABIT) in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Thrasher Research Fund (Other); Emory University (Other)
Responsible Party: Principal Investigator, Andrew Gordon, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08126
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy; Hemiplegia; Children; Pediatric
Keywords: cerebral palsy; constraint-induced therapy; constraint-induced movement therapy; CP; hemiplegia; hand; forced use; motor control; children; HABIT; Hand-arm bimanual intensive therapy; Bilateral training; Bimanual training; functional therapy; physical therapy; occupational therapy; intensive; pediatric; development; upper extremity; hemiplegic
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia; Habits | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIMT Intervention (Experimental): Participants randomized to this arm were provided with 90 minutes of Constraint-Induced Movement Therapy (CIMT), which requires hand restraint and progression of unimanual tasks.
  Interventions: Procedure: Constraint-Induced Movement Therapy (CIMT)
- HABIT Intervention (Experimental): Participants randomized to this arm were provided with 90 minutes of Hand-Arm Bimanual Intensive Therapy (HABIT), which requires that tasks are progressed bimanually.
  Interventions: Procedure: Hand-Arm Bimanual Intensive Therapy (HABIT)

INTERVENTIONS:
Procedure: Constraint-Induced Movement Therapy (CIMT) — 90 hours
  Arms: CIMT Intervention
Procedure: Hand-Arm Bimanual Intensive Therapy (HABIT) — 90 hours
  Arms: HABIT Intervention

SUMMARY:
A randomized control trial of bimanual training. The protocols have been developed at Columbia University to be child friendly and draws upon our experience since 1997 with constraint-induced movement therapy in children with cerebral palsy.

DETAILED DESCRIPTION:
A new treatment involving bimanual (Hand-Arm Bimanual Intensive Therapy (HABIT). The protocols have been developed at Columbia University to be child friendly and draws upon our experience since 1998 with constraint-induced movement therapy in children with cerebral palsy. The interventions are performed in a 15 day day-camp setting with several children and at least one therapist per child. We have conducted 24 day camps to date since 2002, and are now collaborating with clinicians worldwide to expand our treatment availability. The aim is to promote the use of and improve the coordination of movement of both hands together. PARTICIPATION IS FREE. Please check out our website for more information: http://www.tc.edu/centers/cit/.

ELIGIBILITY:
Inclusion Criteria:

willingness to agree to intervention and testing procedures and travel to the University for participation and testing.

Exclusion Criteria:

* health problems not associated with CP
* uncontrollable seizures
* visual problems that would interfere with carrying out the intervention or testing
* botulinum toxin therapy in the upper extremity musculature during the last six months or who wish to receive it within the period of study

Ages: 30 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Gordon, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Background] Charles JR, Wolf SL, Schneider JA, Gordon AM. Efficacy of a child-friendly form of constraint-induced movement therapy in hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2006 Aug;48(8):635-42. doi: 10.1017/S0012162206001356. PMID 16836774
- [Background] Gordon AM, Charles J, Wolf SL. Efficacy of constraint-induced movement therapy on involved upper-extremity use in children with hemiplegic cerebral palsy is not age-dependent. Pediatrics. 2006 Mar;117(3):e363-73. doi: 10.1542/peds.2005-1009. PMID 16510616
- [Background] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Background] Steenbergen B, Charles J, Gordon AM. Fingertip force control during bimanual object lifting in hemiplegic cerebral palsy. Exp Brain Res. 2008 Mar;186(2):191-201. doi: 10.1007/s00221-007-1223-6. Epub 2008 Jan 26. PMID 18224309
- [Background] Schertz M, Gordon AM. Changing the model: a call for a re-examination of intervention approaches and translational research in children with developmental disabilities. Dev Med Child Neurol. 2009 Jan;51(1):6-7. doi: 10.1111/j.1469-8749.2008.03220.x. No abstract available. PMID 19087099
- [Background] Gordon AM, Chinnan A, Gill S, Petra E, Hung YC, Charles J. Both constraint-induced movement therapy and bimanual training lead to improved performance of upper extremity function in children with hemiplegia. Dev Med Child Neurol. 2008 Dec;50(12):957-8. doi: 10.1111/j.1469-8749.2008.03166.x. No abstract available. PMID 19160464
- [Background] Hung YC, Casertano L, Hillman A, Gordon AM. The effect of intensive bimanual training on coordination of the hands in children with congenital hemiplegia. Res Dev Disabil. 2011 Nov-Dec;32(6):2724-31. doi: 10.1016/j.ridd.2011.05.038. Epub 2011 Jun 28. PMID 21715141
- [Result] Gordon AM, Hung YC, Brandao M, Ferre CL, Kuo HC, Friel K, Petra E, Chinnan A, Charles JR. Bimanual training and constraint-induced movement therapy in children with hemiplegic cerebral palsy: a randomized trial. Neurorehabil Neural Repair. 2011 Oct;25(8):692-702. doi: 10.1177/1545968311402508. Epub 2011 Jun 23. PMID 21700924
- See also: Center for cerebral palsy research — http://www.tc.edu/centers/cit/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from clinics in the NYC area, and online support groups from June 2007 to July 2009. Participants were firs screened via e-mail and/or telephone and potentially invited to receive an on-site physical examination or an examination videotaped by their physical occupational therapist.
Groups:
- CIMT: Participants randomized to this arm were provided with 90 minutes of Constraint-Induced Movement Therapy (CIMT), which requires hand restraint and progression of unimanual tasks.
- HABIT: Participants randomized to this arm were provided with 90 minutes of Hand-Arm Bimanual Intensive Therapy (HABIT), which requires that tasks are progressed bimanually.
Period: Overall Study
Arm/Group | CIMT | HABIT
Started | 22 | 22
Completed | 21 | 21
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Failure to complete pretest | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CIMT | HABIT | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (2.2) | 6.4 (1.11) | 6.3 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Assisting Hand Assessment (AHA)
Description: The Assisting Hand Assessment (AHA) quantifies the effectiveness with which a child with unilateral disability uses his/her affected (assisting) hand in bimanual activity. Scores range from 0-100 units, with higher scores signifying better bimanual performance.
Time Frame: Baseline, 6 months
Population: Subject sample size calculation based on prior data. intention to treat (ITT) was used.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | CIMT | HABIT
Number analyzed (Participants) | 21 | 21
score | 0.42 [0.08 to 0.76] | 0.56 [0.23 to 0.90]
Statistical Analysis 1: Comparison: CIMT; ANOVA; Test type: Superiority or Other; p < 0.01, ANOVA — ANOVA; Mean Difference (Final Values) = 1, Standard Deviation 1

2. Primary Outcome: Change in Score on the Jebsen-Taylor Test of Hand Function (JTTHF)
Description: The Jebsen-Taylor Test of Hand Function (JTTHF) is a standardized test of simulated functional tasks quantifying the time to complete a battery of unimanual tasks. The activities performed include flipping index cards, object placement, simulated eating, stacking checkers, and manipulating empty and full cans. Scores range from 0-1080 seconds, with a lower score signifying better hand function.
Time Frame: Baseline, 6 months
Measure: Mean (90% Confidence Interval); unit: score
Arm/Group | CIMT | HABIT
Number analyzed (Participants) | 21 | 21
score | -141.7 [-195.4 to -88.0] | -131.2 [-185.0 to -77.5]

ADVERSE EVENTS:
Arm/Group | CIMT | HABIT
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
Both groups receive treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No